CLINICAL TRIAL: NCT01779050
Title: A Phase II Randomized Trial Evaluating the Effect of Trastuzumab on Disease Free Survival in Early Stage HER2-Negative Breast Cancer Patients With ERBB2 Expressing Bone Marrow Disseminated Tumor Cells
Brief Title: Effect of Trastuzumab on Disease Free Survival in Early Stage HER2-Negative Breast Cancer Patients With ERBB2 Expressing Disseminated Tumor Cells
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Loss of study funding
Sponsor: Washington University School of Medicine (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201309084
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Results first posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Trastuzumab; Cyclophosphamide; carboxypeptidase M; Paclitaxel; Albumin-Bound Paclitaxel; Epirubicin; Docetaxel; Carboplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (definitive therapy) (Active Comparator): Patients receive definitive surgery and best practice standard chemotherapy according to NCCN guidelines. The 5 chemo backbone options are:
  * doxorubicin or epirubicin plus cyclophosphamide followed by paclitaxel or docetaxel
  * docetaxel plus cyclophosphamide
  * single-agent paclitaxel
  * docetaxel plus carboplatin
  * fluorouracil plus epirubicin plus cyclophosphamide followed by paclitaxel or docetaxel
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Paclitaxel; Drug: Epirubicin; Drug: Docetaxel; Drug: Fluorouracil
- Arm II (definitive therapy, trastuzumab) (Experimental): Patients receive definitive surgery and best practice standard chemotherapy according to NCCN guidelines. The 5 chemo backbone options are:
  * doxorubicin or epirubicin plus cyclophosphamide followed by paclitaxel or docetaxel
  * docetaxel plus cyclophosphamide
  * single-agent paclitaxel
  * docetaxel plus carboplatin
  * fluorouracil plus epirubicin plus cyclophosphamide followed by paclitaxel or docetaxel
  Patients will also receive trastuzumab IV over 30-90 minutes for 52 weeks starting such that there is a minimum of 8 weeks of overlap with the standard of care chemotherapy. Trastuzumab may be given weekly, every 2 weeks, or every 3 weeks while overlapping with standard of care chemotherapy. Trastuzumab will be given every 3 weeks after all standard of care chemotherapy has concluded. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Doxorubicin; Biological: Trastuzumab; Drug: Cyclophosphamide; Drug: Paclitaxel; Drug: Epirubicin; Drug: Docetaxel; Drug: Carboplatin; Drug: Fluorouracil

INTERVENTIONS:
Drug: Doxorubicin
  Other Names: Adriamycin®, Rubex®, Hydroxydaunomycin Hydrochloride, Hydroxydoxorubicin Hydrochloride
Biological: Trastuzumab
  Other Names: •Herceptin®
  Arms: Arm II (definitive therapy, trastuzumab)
Drug: Cyclophosphamide
  Other Names: Cytoxan®, CPM, CTX, CYT
Drug: Paclitaxel
  Other Names: Abraxane®, Onxol®
Drug: Epirubicin
  Other Names: Ellence, Pharmorubicin, Epirubicin ebewe
Drug: Docetaxel
  Other Names: Taxotere, Docefrez
Drug: Carboplatin
  Other Names: cis-Diammine(1,1-cyclobutanedicarboxylato)platinum(II), Paraplatin, Paraplatin-AQ
  Arms: Arm II (definitive therapy, trastuzumab)
Drug: Fluorouracil
  Other Names: 5-FU, Adrucil

SUMMARY:
This phase II trial studies the efficacy of trastuzumab treatment in breast cancer patients with stage II-III human epidermal growth factor receptor 2 (HER2)-negative tumors and HER2-expressing bone marrow disseminated tumor cells (DTCs). Administering targeted trastuzumab therapy to these patients may result in the elimination of HER2 expressing disseminated tumor cells and improved disease free survival.

ELIGIBILITY:
Pre-Registration Inclusion Criteria:

* Histologically confirmed HER2-negative primary invasive ductal or invasive lobular breast carcinoma. For patients enrolling for neoadjuvant treatment, diagnosis must be clinical stage II or III; for patients enrolling for adjuvant treatment, diagnosis must be pathologic stage IIA to IIIC. Standard HER2 testing will be performed in the surgical specimen at Washington University according to the standard of care in the Department of Pathology. A HER2-negative primary breast cancer sample from a patient eligible for randomization should have a HER2 IHC score of 0 or 1+ Those patients with IHC score of 2+ should be HER2 FISH-negative in standard testing. Patient will have undergone staging studies including a CT of the chest/abdomen/pelvis and bone scan and/or PET scan either prior to the initiation of treatment or prior to entry into the trial. In addition, patients with non-metastatic, HER2-negative, recurrent tumors who need chemotherapy are eligible.
* Planning to receive best practice adjuvant or neoadjuvant chemotherapy according to institutional guidelines. Adjuvant tamoxifen or aromatase inhibitors treatment will be allowed for hormone receptor-positive patients. Patients who have failed neoadjuvant endocrine therapy will also be eligible.
* At least 18 years old.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
* Patient (or legally authorized representative) must be able to understand and willing to sign a written informed consent document.

Pre-Registration Exclusion Criteria:

* Prior chemotherapy for this cancer (excluding initiation of best practice chemotherapy to be given as standard of care as described in this protocol, which may be initiated after the pre-registration bone marrow collection but before final confirmation of eligibility and randomization).
* Previous treatment with trastuzumab or any other Her2 targeted therapy.
* Presence of an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Registration Inclusion Criteria

* Presence of bone marrow ERBB2 overexpressing DTCs at the time of diagnosis; bone marrow aspiration will be performed in consented patients to evaluate DTCs following pre-registration provided patients meet all eligibility criteria as described in this section.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
* Adequate cardiac function as demonstrated by LVEF of >55% performed no more than 4 weeks prior to randomization.
* Normal organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * hemoglobin ≥ 10 g/dL
  * total bilirubin within institutional upper limits of normal unless related to primary disease
  * AST(SGOT)/ALT(SGPT) ≤2.0 X institutional upper limit of normal
  * Creatinine ≤ 1.5 institutional upper limits of normal OR creatinine clearance ≥60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* If a woman of childbearing potential, patient must use two forms of effective contraception for a minimum of 6 months following trastuzumab. Effective methods of birth control include use of established oral, injected, or implanted hormonal methods of birth control, IUD, IUS, and condoms.

Registration Exclusion Criteria

* Evidence of distant metastasis present by CT scan, bone scan, or physical exam.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to trastuzumab.
* Prior chemotherapy for this cancer (excluding initiation of best practice chemotherapy to be given as standard of care described in this protocol, which may be initiated after the pre-registration bone marrow collection but before final confirmation of eligibility and randomization).
* History of other malignancy ≤ 5 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Pregnant or breastfeeding. Patient must have a negative serum pregnancy test ≤ 7 days from date of registration (if a woman of childbearing potential).
* Clinically important history of active liver disease, including viral or other hepatitis or cirrhosis.
* Uncontrolled hypocalcemia, hypomagnesemia, hyponatremia, or hypokalemia defined as less than the lower limit of normal for the institution despite adequate electrolyte supplementation.
* Symptomatic intrinsic lung disease or extensive tumor involvement of the lungs resulting in dyspnea at rest.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-12-19 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Aft, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siddappa CM, Watson MA, Pillai SG, Trinkaus K, Fleming T, Aft R. Detection of disseminated tumor cells in the bone marrow of breast cancer patients using multiplex gene expression measurements identifies new therapeutic targets in patients at high risk for the development of metastatic disease. Breast Cancer Res Treat. 2013 Jan;137(1):45-56. doi: 10.1007/s10549-012-2279-y. Epub 2012 Nov 6. PMID 23129172
- [Background] Rack B, Juckstock J, Gunthner-Biller M, Andergassen U, Neugebauer J, Hepp P, Schoberth A, Mayr D, Zwingers T, Schindlbeck C, Friese K, Janni W. Trastuzumab clears HER2/neu-positive isolated tumor cells from bone marrow in primary breast cancer patients. Arch Gynecol Obstet. 2012 Feb;285(2):485-92. doi: 10.1007/s00404-011-1954-2. Epub 2011 Jun 30. PMID 21717141
- [Background] Vincent-Salomon A, Pierga JY, Couturier J, d'Enghien CD, Nos C, Sigal-Zafrani B, Lae M, Freneaux P, Dieras V, Thiery JP, Sastre-Garau X. HER2 status of bone marrow micrometastasis and their corresponding primary tumours in a pilot study of 27 cases: a possible tool for anti-HER2 therapy management? Br J Cancer. 2007 Feb 26;96(4):654-9. doi: 10.1038/sj.bjc.6603584. Epub 2007 Jan 30. PMID 17262082
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Definitive Therapy) | Arm II (Definitive Therapy, Trastuzumab)
Started | 4 | 3
Completed | 3 | 3
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Definitive Therapy) | Arm II (Definitive Therapy, Trastuzumab) | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Median (Full Range); unit: years] | 63.5 [54 to 75] | 58 [55 to 74] | 63 [54 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Disease Recurrence
Description: -Disease recurrence is defined as the documented appearance of local (breast, chest wall, axillary, supraclavicular nodes) or distant disease.
Time Frame: Up to 3 years after completion of treatment (estimated to be 4 years)
Population: One participant in Arm 1 was not evaluable as they withdrew before receiving any treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Definitive Therapy) | Arm II (Definitive Therapy, Trastuzumab)
Number analyzed (Participants) | 3 | 3
Participants | 1 | 0

2. Primary Outcome: Death Rate
Time Frame: Up to 3 years after completion of treatment (estimated to be 4 years)
Population: One participant in Arm 1 was not evaluable as they withdrew before receiving any treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Definitive Therapy) | Arm II (Definitive Therapy, Trastuzumab)
Number analyzed (Participants) | 3 | 3
Participants | 1 | 0

3. Secondary Outcome: Elimination of ERBB2 Overexpressing Bone Marrow DTCs
Description: Bone marrow disseminated tumor cells (DTCs) are evaluated by RT-PCR performed on specimens collected 6-18 months apart (one before and one after therapy). The proportion of samples turned negative after therapy will be calculated. Samples will be considered negative for ERBB2-expression if expression from bone marrow collected from each iliac crest is less than 2 standard deviations above the ERBB2-level in pooled normal bone marrow specimens.
Time Frame: Before treatment and after treatment (estimated to be 6-18 months)
Population: Data was not collected.
Arm/Group | Arm I (Definitive Therapy) | Arm II (Definitive Therapy, Trastuzumab)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: -Adverse events were collected from the time informed consent was obtained and initiation of study procedures and ended 30 days following the last day of study treatment or study discontinuation/termination, whichever was earlier. Median length of follow-up for adverse event data was 272 days (full range 135 days-395 days). -All-cause mortality was assessed for up to 4 years.
Arm/Group | Arm I (Definitive Therapy) | Arm II (Definitive Therapy, Trastuzumab)
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Definitive Therapy) (N=3) | Arm II (Definitive Therapy, Trastuzumab) (N=3)
Decreased LVEF-asymptomatic (Cardiac disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 3
Dry mouth (Gastrointestinal disorders) | 2 | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1
Edema limbs (General disorders) | 0 | 2
Fatigue (General disorders) | 3 | 3
Fever (General disorders) | 2 | 1
Nasal mucosal infection (Infections and infestations) | 1 | 0
Shingles (Infections and infestations) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Bruising to arms and legs (Injury, poisoning and procedural complications) | 0 | 1
Hemoglobin increased (Investigations) | 0 | 1
Neutropenia (Investigations) | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain-left side (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 3
Lethargy (Nervous system disorders) | 2 | 1
Neuropathy - sensory (Nervous system disorders) | 2 | 1
Tremors (Nervous system disorders) | 0 | 1
Amnesia (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 2
Depression (Psychiatric disorders) | 3 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Breast enlargement (post-radiation change) (Reproductive system and breast disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Weeping rash beneath breast (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 2
Atrophy (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Left pointer finger laceration (Skin and subcutaneous tissue disorders) | 0 | 2
Nail loss (Skin and subcutaneous tissue disorders) | 1 | 1
Nonhealing left leg sore (Skin and subcutaneous tissue disorders) | 0 | 1
Hot flashes (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT01779050/Prot_SAP_000.pdf